CLINICAL TRIAL: NCT04066660
Title: Study of Oligo-Fucoidan in Advanced Hepatocellular Carcinoma (HCC)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: After interim analysis, we planned to recruit 100 participants. However, due to COVID-19 challenges, statistician advised each group needs at least 30 samples (Gay, 1992). The sponsor and team decided to terminate the trial early for valid data.
Sponsor: Hi-Q Marine Biotech International, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HiQ-FUCO-003
Record Dates: First submitted 2019-08-20; First posted 2019-08-26 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: Oligo Fucoidan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment & Oligo Fucoidan (Experimental): 4.4 g Oligo Fucoidan powder by six months, BID
  Interventions: Dietary Supplement: Oligo Fucoidan
- Treatment & Placebo (Placebo Comparator): 4.4 g Placebo powder by six months, BID
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Oligo Fucoidan — 4.4 g oligo fucoidan powder, oral, BID
  Arms: Treatment & Oligo Fucoidan
Dietary Supplement: Placebo — 4.4 g placebo powder, oral, BID
  Arms: Treatment & Placebo

SUMMARY:
A randomized, double-blind, controlled trial was conducted evaluating the efficacy of Oligo-Fucoidan with the molecular weight ranged from 500 to 800 Da. as a supplemental therapy in patients with advanced hepatocellular carcinoma. The previous study results demonstrate the advantages of Oligo-Fucoidan in improving the disease control rate in metastatic colorectal cancer. The previous study might provide insights into the development of cancer treatments, particularly in the combination of natural or herbal products with chemotarget agents.

DETAILED DESCRIPTION:
Oligo-Fucoidan, a heparin-like molecule with high percentages of L-fucose and sulfated ester groups and low percentages of D-xylose, D-galactose, D-mannose, and glucuronic acid, was present in the cell wall matrix of brown seaweed. Brown seaweed Oligo-Fucoidan was reported to demonstrate various biological activities such as antioxidant, anti-inflammatory, antiproliferative, and proapoptotic activities. Oligo-Fucoidan was also revealed to inhibit the growth of breast and lung cancers in animal models. Oligo-Fucoidan treatment induces the degradation of transforming growth factor (TGF)-β receptor and the consequent inhibition of the epithelial-mesenchymal transition (EMT) in cancer cells. In addition to these molecular mechanisms, it is imperative to investigate the potential of Oligo-Fucoidan as a miRNA regulator for breast cancer treatment and thus delineate the molecular mechanisms underlying the anticancer effects of Oligo-Fucoidan. A randomized, double-blind, controlled trial was conducted evaluating the efficacy of Oligo-Fucoidan with the molecular weight ranged from 500 to 800 Da. as a supplemental therapy in patients with . advanced hepatocellular carcinoma. The previous study results demonstrate the advantages of Oligo-Fucoidan in improving the disease control rate in metastatic colorectal cancer. The previous study might provide insights into the development of cancer treatments, particularly in the combination of natural or herbal products with chemotarget agents.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years;
* ECOG PS 0-2;
* Histologically or cytologically documented unresectable HCC;
* Measurable disease by RECIST criteria;
* HCC without well control
* Child-Pugh A-B
* Albumin ≥ 2.8 g/dl;
* Serum total bilirubin ≤ 3 mg/dl;
* INR ≤ 2.3 or PT ≤ 6 seconds above control;
* WBC ≥ 2,500/µl;
* ANC ≥ 1,000/µl;
* Platelets ≥ 50,000/µl;
* Hb ≥ 8.5 g/dl;
* Creatinine ≤ 1.5 x ULN; AND

Exclusion Criteria:

* Metastatic tumors;
* Prior or concomitant systemic anti-cancer treatment for HCC, including:
* Systemic chemotherapy (TACE is allowed)
* Investigational anti-cancer agents
* Severe and/or uncontrolled medical conditions:
* Uncontrolled high blood pressure
* History of poor compliance with anti-hypertensive agents
* Active or uncontrolled infection
* Unstable angina
* CHF
* MI or CVA < 6 months
* GI bleeding < 30 days
* Unable to take oral medications
* Severe renal impairment which requires dialysis; proteinuria > grade 2;
* BMT or stem cell rescue < 4 months; organ transplant;
* HIV infection;
* Major surgical procedure, open biopsy, or significant traumatic injury < 4 weeks or those who receive minor surgical procedures (e.g. core biopsy or fine needle aspiration) within 2 weeks;
* Patients taking narrow therapeutic index medications will be monitored closely. These include warfarin, phenytoin, quinidine, carbamazepine, phenobarbital, cyclosporine, and digoxin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Disease Control Rate | from Day 1 to end of treatment (4th visit, month 6)
  Disease Control Rate will be evaluated by mRECIST

SECONDARY OUTCOMES:
Objective Response Rate | Screening (baseline), complete of Treatment Phase(month 6)
  Objective Response Rate will be evaluated using measurements according to mRECIST
Quality of Life (QoL) | 1st visit to 4th visit (from day 1 to month 6)
  Quality of Life will be evaluated by questionnaire based on EORTC-QLQ30, specific questions evaluated by scores from 1 (not at all), 2 (a little), 3 (quite a bit), 4 (very much); overall healthy and quality of life will be evalauted by scores from 1 (very poor) to 7 (excellent)

CONTACTS AND LOCATIONS:
Overall Officials: Xizhong Shen, PhD, Study Director — Shanghai Zhongshan Hospital
Locations (1):
- Fudan University Zhongshan Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No